CLINICAL TRIAL: NCT06414122
Title: The Efficacy of Modulated Mid-frequency (Whole-body Electromyostimulation) and Nutritional Therapy in Patients With Solid Tumors of the Gastrointestinal Tract (Excluding Liver and Pancreatic Carcinomas)
Brief Title: Modulated Mid-frequency Whole-body Electromyostimulation and Nutritional Therapy in Gastrointestinal Cancer Patients
Acronym: MOMENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Helen Schörghofer, Helen Schörghofer, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-1294
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Oesophageal Cancer; Gastric Cancer; Duodenal Cancer; Colorectal Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Duodenal Neoplasms; Colorectal Neoplasms | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WB-EMS (Experimental): Intervention group receives multimodal therapy with whole-body electromyostimulation and exercise therapy (WB-EMS) as well as conventional nutritional counseling with guidelines and digital nutritional coaching
  Interventions: Other: mid-frequency whole-body electromyostimulation (WB-EMS); Other: nutritional therapy
- CONTROL (Active Comparator): Control group receives multimodal therapy with moderate conventional exercise training in a group and conventional nutritional counselling with guidelines and digital nutritional coaching
  Interventions: Other: conventional exercise training; Other: nutritional therapy

INTERVENTIONS:
Other: mid-frequency whole-body electromyostimulation (WB-EMS) — supervised group training sessions at least once and optionally twice a week, lasting 11-20 minutes, over 12 weeks, 12-24 training sessions in total
  Arms: WB-EMS
Other: conventional exercise training — supervised group training at least once a week, optional additional home-based training once a week, lasting 40 minutes, over 12 weeks, 12-24 training sessions in total
  Arms: CONTROL
Other: nutritional therapy — conventional nutritional counselling with guidelines and digital nutritional coaching

SUMMARY:
The purpose of this study is to assess the efficacy of modulated mid-frequency whole-body electromyostimulation (WB-EMS) combined with nutritional therapy in patients with gastrointestinal cancer.

DETAILED DESCRIPTION:
This study aims to combine the applicability and effectiveness of a form of strength training with targeted nutritional training. For this purpose, training with electromyostimulation (application of modulated mid-frequency; WB-EMS) is carried out, which pursues the effect of cell activation and the improvement of muscle strength. The primary aim of the multimodal intervention presented here is to increase muscle mass and improve energy utilisation and metabolism. Patients should experience increased mobility and independence as a result of this intervention. In the study, patients are randomly assigned to one of two groups, with one group receiving an application of electricity and the other group performing standardised exercise therapy without electricity. Otherwise, the groups do not differ in the applications or tests. In addition, nutritional coaching takes place in both groups with digital nutritional coaching.

Patients with a malignant tumour of the oesophagus, stomach, duodenum or colon or rectum with medical therapy administered before or after surgery (neoadjuvant and adjuvant therapy) and after surgery without further therapy can participate in the study.

The aim is to compare the use of electromyostimulation in this multimodal approach regarding its effectiveness in terms of muscle growth compared to the conventional multimodal approach. The research hypothesis is that the additional training stimulus provided by the application of electricity leads to significantly higher muscle growth than conventional training without electricity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oesophageal, gastric, duodenal, colon or rectal cancer following surgery without further therapy and with neoadjuvant and adjuvant therapy
* medical clearance for exercise training
* written declaration of consent from the study participant

Exclusion Criteria:

* Participation in another study on the topic of exercise or nutrition
* Electronic implants such as pacemakers, pumps, and coronary stents
* Cardiac arrhythmia
* Implants in the area of application (e.g. breast implants)
* Pregnancy
* Epilepsy
* Wounds and open skin diseases in the area of application of the electrodes
* Unhealed operations or bone fractures
* Acute inflammatory diseases (e.g. inflammation of the intervertebral discs, bones, vessels, or soft tissue)
* Directly after herniated discs or other instabilities such as large abdominal wall hernias
* Blood clots (thromboses)
* Bone diseases with high-grade osteoporosis
* Increased risk of haemorrhage
* Fever and illnesses that can be aggravated by physical exertion
* Untreated high blood pressure
* Blindness
* Continuous parenteral nutrition
* Metal and electronic parts in the body (e.g. prostheses, metal vascular clips, hearing aids/inner ear/cochlear implants, magnetic dental prostheses, pacemakers, contraceptives)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Muscle mass of the quadriceps muscle | Baseline and week 12
  Muscle mass of the quadriceps muscle (vastus lateralis / rectus femoris), cross-sectional diameter (CSD) using ultrasound. Muscle ultrasound represents a cheap and user-friendly, yet robust and reliable, method to monitor muscle mass.

SECONDARY OUTCOMES:
Body composition | Baseline and week 12
  Body composition including skeletal muscle mass, fat free mass, fat mass, total body water, body cell mass and extracellular mass, using bioimpedance analysis (BIA) (Nutriguard-MS)
Performance Status | Baseline and week 12
  Performance Status, with the help of Karnofsky Index (range 0 - 100, higher = better)
Endurance capacity | Baseline and week 12
  Endurance capacity, using spiroergometry measuring maximal oxygen uptake (VO2 max) (higher = better)
Lower limb performance | Baseline and week 12
  Lower limb performance, using 1 minute sit-to-stand test (higher = better)
Upper limb performance | Baseline and week 12
  Upper limb performance, using hand grip strength dynamometry (higher = better)
Fatigue | Baseline and week 12
  Fatigue symptoms, using the 13-item Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT Fatigue Scale). The FACIT-Fatigue is a 13-item measure that assesses self-reported fatigue and its impact on daily activities and function. Score range 0-52 (higher = better)
health-related Quality of life | Baseline and week 12
  Quality of life, using the EORTC QLG Core Questionnaire (EORTC QLQ-C30). The EORTC QLQ-C30 is a 30-item instrument meant to assess some of the different aspects that define the quality of life of cancer patients. Score range 0-100 (higher = better)

CONTACTS AND LOCATIONS:
Overall Officials: Freerk T Baumann, Univ.-Prof., Principal Investigator — Universitätsklinikum Köln
Locations (1):
- Universitätsklinikum Köln, Centrum für Integrierte Onkologie (CIO), Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Time Frame: Beginning 6 months and ending 24 months after article publication
Access Criteria: IPD will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to helen.schoerghofer@uk-koeln.de. To gain access, data requestors will need to sign a data access agreement.